CLINICAL TRIAL: NCT00337129
Title: Phase II Evaluation of E7389 (NSC-707389) in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: S0618 E7389 in Treating Patients With Metastatic or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03046; U10CA032102 (NIH); S0618 (Other: SWOG); CDR0000481530 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
Keywords: metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eribulin mesylate (Experimental): eribulin mesylate
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — 1.4 mg/m2 by IV bolus on Days 1 and 8 of an every 21-day cycle.
  Other Names: E7389

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as E7389, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well E7389 works in treating patients with metastatic or recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the response probability (confirmed, complete, and partial responses) in patients with metastatic or recurrent squamous cell carcinoma of the head and neck treated with E7389.
* Estimate progression-free and overall survival probability in these patients.
* Evaluate the qualitative and quantitative toxicities of this treatment regimen.

OUTLINE: This is a multicenter study.

Patients receive E7389 IV on days 1 and 8. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (SCCHN)

  * Disease is either metastatic at diagnosis or has persisted, metastasized, or recurred after definitive surgery and/or radiotherapy
  * Not amenable to surgical resection for salvage therapy
  * No newly diagnosed nonmetastatic disease
  * No salivary or nasopharyngeal primary disease
  * Patients who have failed primary surgery alone, and who have disease that is salvageable by radiation or chemoradiation, are not eligible
* Measurable disease

  * Measurable disease within a previous radiotherapy port must demonstrate clearly progressive disease
* No active or prior CNS metastasis

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2 times ULN
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known HIV positivity
* No prior malignancies except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer currently in complete remission
  * Any other cancer for which the patient has been disease free for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for recurrent or newly diagnosed metastatic disease
* At least 6 months since prior induction or adjuvant chemotherapy for patients who relapsed after receiving this therapy

  * No more than 1 prior induction or adjuvant regimen (may have included a taxane)
* More than 2 weeks since prior biologic therapy (i.e., epidermal growth factor inhibitors and vascular endothelial growth factor inhibitors)
* More than 28 days since prior radiotherapy and recovered
* More than 28 days since prior surgery and recovered
* No other concurrent therapy (i.e., radiotherapy, chemotherapy, immunotherapy, biologic therapy, or gene therapy) for SCCHN
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent prophylactic colony-stimulating factors during course 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M. Arnold, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky
Locations (139):
- United States (139):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2006 to December, 2007 a total of 42 patients were enrolled from SWOG institutions
Pre-assignment Details: 2 patients are not eligible before assignment.
Groups:
- Treatment (E7389 IV): Patients receive E7389 IV on days 1 and 8 of an every 21-day cycle.
Period: Overall Study
Arm/Group | Treatment (E7389 IV)
Started | 40
Completed | 0 (Treatment is not for a fixed period and continues until discontinuation criterion is met.)
Not Completed | 40
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 32
Not completed — Death | 2
Not completed — not protocol specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (E7389 IV)
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Probability (Confirmed Complete and Partial Responses)
Description: Response was defined per RECIST. Complete response (CR) was defined as complete disappearance of all baseline measurable and non-measurable disease with no new lesions. Partial response (PR) was defined as at least 30% decrease under baseline of the sum of longest diameters of all target measurable lesions with no unequivocal progression of non-measurable disease and no new lesions. A CR or PR must be confirmed by a second determination at least 4 weeks apart. All disease must have been assessed using the same technique as baseline.
Time Frame: Every 6 weeks until progression of disease up to a maximum of 3 years after registration
Population: Only eligible patients were included in the analysis
Measure: Number; unit: participants
Arm/Group | Treatment (E7389 IV)
Number analyzed (Participants) | 40
participants
  Complete Response | 0
  Partial Response | 2
  No Response | 38
Statistical Analysis 1: Comparison: Treatment (E7389 IV); Null hypothesis: response probability < 5%; alternative hypothesis: response probability > 20%. A two-stage design was used. If no responses among the first 20 patients, the study would be terminated with the conclusion that E7389 is inactive. However, if at least one response was seen then an additional 20 patients would be accrued. Five or more responses out of 40 would be considered evidence that E7389 warranted further study. This design had a significance level of 5% and a power of 92%; Test type: Superiority or Other; two-stage binomial; Response probability = 0.05, 95% CI 2-sided [0.01 to 0.17]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from date of registration to the date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at date of last contact.
Time Frame: Every 6 weeks until progression of disease up to a maximum of 3 years after registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (E7389 IV)
Number analyzed (Participants) | 40
months | 3 [1 to 3]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of registration to the date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Every 3 months for first year, then every six months thereafter up to a maximum of 3 years from registration.
Population: Only eligible patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (E7389 IV)
Number analyzed (Participants) | 40
months | 7 [5 to 10]

4. Secondary Outcome: Participants With a Given Type of AE
Description: The NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0 was utilized.
Time Frame: Every 3 weeks while on protocol therapy, up to 3 years.
Population: All eligible patients who started protocol treatment are included in analysis of toxicity
Measure: Number; unit: participants
Arm/Group | Treatment (E7389 IV)
Number analyzed (Participants) | 40
participants
  Dehydration | 1
  Diarrhea | 2
  Dry mouth/salivary gland (xerostomia) | 1
  Dyspnea (shortness of breath) | 2
  Fatigue (asthenia, lethargy, malaise) | 2
  Glucose, serum-high (hyperglycemia) | 1
  Hemoglobin | 1
  Hemorrhage - Bronchopulmonary NOS | 1
  Infection w/ Grade 3/4 ANC - Skin (cellulitis) | 1
  Infection w unk ANC - gums (gingivitis) | 1
  Leukocytes (total WBC) | 5
  Lymphopenia | 6
  Mucositis - gums (gingivitis) | 1
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 4
  Pneumonitis/pulmonary infiltrates | 1
  Potassium, serum-low (hypokalemia) | 1
  Sodium, serum-low (hyponatremia) | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed on Day 1 and Day 8 of every 21-day cycle of treatment.
Description: This study utilized the CTCAE (NCI Common Toxicity Criteria for Adverse Events) version 3.0
Groups:
- Treatment (E7389 IV): Patients receive E7389 IV on days 1 and 8 of an every 21-day cycle. Includes only patients who received drug.
Arm/Group | Treatment (E7389 IV)
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (E7389 IV) (N=40)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Infection (documented clinically or microbiologically) with Grade3 or 4 neutrophils-Skin(cellulitis) (Infections and infestations) | 1
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Weight loss (Investigations) | 1
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (E7389 IV) (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 20
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 9
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Pain - Oral cavity (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Oral cavity-gums (gingivitis) (Infections and infestations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 4
Alkaline phosphatase (Investigations) | 5
Leukocytes (total WBC) (Investigations) | 11
Lymphopenia (Investigations) | 9
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 12
Platelets (Investigations) | 2
Weight loss (Investigations) | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 5
Pain - Head/headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less